CLINICAL TRIAL: NCT05701306
Title: A Phase I Clinical Study of APG-115 Alone or in Combination With APG-2575 in Children With Recurrent or Refractory Neuroblastoma or Solid Tumors
Brief Title: APG-115 Alone or in Combination With APG-2575 in Children With Recurrent or Refractory Neuroblastoma or Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: Suzhou Yasheng Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APG115XC103
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Neuroblastoma; Solid Tumor
Keywords: Neuroblastoma; Solid Tumor; APG-115
MeSH Terms: conditions — Neuroblastoma | interventions — Lisaftoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APG-115 monotherapy in part1 (Experimental): Multiple dose cohorts, to determine the RP2D of APG-115.
  Interventions: Drug: APG-115
- APG-115 combined with APG-2575 in part2 (Experimental): Multiple dose cohorts of APG-2575, to determine the RP2D of APG-2575 combined with APG-115.
  Interventions: Drug: APG-115; Drug: APG-2575

INTERVENTIONS:
Drug: APG-115 — Orally once every other day(QOD) for 2 weeks and suspended for 1 week, 21 days as a cycle.
Drug: APG-2575 — Orally once a day (QD) for 21 days, 21 days as a cycle.
  Arms: APG-115 combined with APG-2575 in part2

SUMMARY:
An open, non-randomized Phase I trial of dose-escalation and cohorts expansion to evaluate the safety, pharmacokinetic profile and initial efficacy of APG-115 alone or in combination with APG-2575 in the treatment of recurrent or refractory pediatric neuroblastoma or solid tumors.

DETAILED DESCRIPTION:
Part 1: Dose escalation and expansion of APG-115 monotherapy in pediatric neuroblastoma or solid tumors to determine MTD and recommended phase 2 dose, RP2D.

Part 2: Dose escalation of APG-2575 to determine the MTD and RP2D combined with APG-115 at the dose level determined in part 1 in pediatric neuroblastoma or solid tumor, and extend the RP2D level of the combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent or refractory neuroblastoma or solid tumor.
2. Physical state score ≥ 50.
3. Expected survival ≥ 3 months.
4. There are target lesions (neuroblastoma) or measurable lesions (other solid tumors).
5. Have adequate organ function.
6. Fresh or archived tumor tissue samples should be provided prior to treatment. If none of these specimens are available, inclusion may be made after consultation with the sponsor.
7. Fertile women (≥14 years of age or having menarche) must have a negative serum pregnancy test at the time of the screening visit and must not be breastfeeding or planning to become pregnant during the study period.
8. A potentially fertile male subject (who has spermatoses) or female subject (ibid.) must agree to use effective contraception during the trial period and for 3 months after the trial ends (or is prematurely discontinued).
9. Informed consent must be obtained before carrying out any study procedure specified in the test. For child subjects, the consent of the subject and one of the parent/legal guardian must be obtained.
10. The ability to swallow research drugs.

Exclusion Criteria:

1. Systemic antitumor therapy, including biotherapy, chemotherapy, surgery, radiotherapy, immunotherapy, and other investigational drug therapy (other than placebo), was received within 21 days prior to the first treatment with the study drug.
2. Small-molecule targeted drug therapy was administered 14 days before the first treatment of the study drug or within a known five-half-life period, whichever is shorter.
3. Patients who, according to the investigators' judgment, did not recover sufficiently after surgical treatment. Patients who underwent major surgery within 28 days before receiving the study drug for the first time.
4. Adverse events due to previous antitumor therapy (except grade 2 peripheral neurotoxicity and alopecia that the investigators judged to be of no safety risk) have not recovered (severity higher than grade 1 according to CTCAE version 5.0).
5. Patients with active brain tumors or brain metastases.
6. Active gastrointestinal diseases (e.g. Crohn's disease, ulcerative colitis, or short bowel syndrome) or other malabsorption syndromes that may affect drug absorption.
7. A known hemorrhagic predisposition/disease, such as a history of non-chemotherapy-induced thrombocytopenic bleeding within 1 year before first receiving the study drug; Have active immune thrombocytopenic purpura (ITP), active autoimmune hemolytic anemia (AIHA), or a history of platelet transfusion failure (within 1 year before first receiving the study drug); Severe gastrointestinal bleeding occurred within 3 months.
8. Clinically significant cardiovascular disease, cardiomyopathy, myocardial infarction or history within 6 months prior to administration.
9. Symptomatic active fungal, bacterial, and/or viral infections requiring systemic treatment.
10. Unexplained fever > 38.5℃ within 2 weeks prior to initial administration (subjects with tumor-related fever, as determined by the investigator, could be enrolled).
11. Received MDM2 inhibitors or BCL-2 inhibitors.
12. Any other circumstances or conditions that the investigator considers the patient inappropriate for participation in the study.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (Phase I) | Up to 21 days
  DLT will be defined based on the rate of drug-related grade 3-5 adverse events experienced within the first 3 weeks of study treatment. These will be assessed via CTCAE version 5.0.
Treatment-Emergent Adverse Events per NCI-CTCAE version 5.0 | Up to 12 months
  Number of patients with adverse event; Number of patients with abnormal vital signs, abnorma physical examination, laboratory abnormalities, and abnormal 12-lead ECG in monotherapy of APG-115 and combined with APG-2575.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Tongji Hospital, Huazhong University of Science and Technology (HUST), Wuhan, Hubei
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality